CLINICAL TRIAL: NCT02028104
Title: Open Label Study of Autologous Bone Marrow Mononuclear Cells in Traumatic Brain Injury
Brief Title: Stem Cell Therapy in Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-06
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cells (Experimental): autologous bone marrow mononuclear cell transplantation
  Interventions: Biological: Autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Biological: Autologous bone marrow mononuclear cell transplantation — bone marrow derived mononuclear cells are administered intrathecally in traumatic brain injury patients

SUMMARY:
The purpose of this study was to study the effect of stem cell therapy on common symptoms in patients with Traumatic Brain Injury

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of chronic traumatic brain injury
* Age above 6 months

Exclusion Criteria:

* presence of acute infections such as Human immunodeficiency virus/Hepatitis B - Virus/Hepatitis C Virus
* malignancies
* bleeding tendencies
* pneumonia
* renal failure
* severe liver dysfunction
* severe anemia [Hemoglobin < 8]
* any bone marrow disorder
* space occupying lesion in brain
* other acute medical conditions such as respiratory infection and pyrexia
* pregnancy
* lactation

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in clinical symptoms of traumatic brain injury | 6 months

SECONDARY OUTCOMES:
Disability Rating scale | 6 months

OTHER OUTCOMES:
SF-8 scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alok K Sharma, M.S., M.Ch, Principal Investigator — Neurogen Brain and Spine Institute
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DH, Lee JY, Oh BM, Phi JH, Kim SK, Bang MS, Kim SU, Wang KC. Functional recovery after injury of motor cortex in rats: effects of rehabilitation and stem cell transplantation in a traumatic brain injury model of cortical resection. Childs Nerv Syst. 2013 Mar;29(3):403-11. doi: 10.1007/s00381-012-1969-4. Epub 2012 Nov 24. PMID 23180314
- [Background] Tian C, Wang X, Wang X, Wang L, Wang X, Wu S, Wan Z. Autologous bone marrow mesenchymal stem cell therapy in the subacute stage of traumatic brain injury by lumbar puncture. Exp Clin Transplant. 2013 Apr;11(2):176-81. doi: 10.6002/ect.2012.0053. Epub 2012 Aug 11. PMID 22891928